CLINICAL TRIAL: NCT01851928
Title: The Validation of Two Inpatient Adult Nutrition Screening Tools in Cancer Care - a Prospective Study
Brief Title: Validation of a Nutrition Screening Tool
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 3621
Record Dates: First submitted 2012-04-20; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Cervical Cancer; Endometrial Cancer; Esophageal Cancer; Fallopian Tube Cancer; Gastric Cancer; Ovarian Cancer; Sarcoma; Vaginal Cancer; Vulvar Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Fallopian Tube Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to evaluate the sensitivity and specificity of two nutrition screening tools to identify inpatients with malnutrition or at risk of malnutrition. The two tools are the Royal Marsden Abridged Adult Nutrition Screening Tool (AANST) and the Malnutrition Screening Tool (MST)[10] The tools will be compared with the currently accepted gold standard, Patient Generated Subjective Global Assessment (PG-SGA). Both screening tools are in the form of scored questionnaires and are suitable for electronic input.

The ultimate objective is to select an adult inpatient nutrition screening tool with the highest sensitivity for future use in the oncology inpatient setting in order to allow prompt commencement of an appropriate nutrition care plan.

ELIGIBILITY:
Inclusion Criteria:

* All adult inpatients, over the age of 18, admitted to RMH for whom a measured weight and height can be obtained

Exclusion Criteria

* Patients for whom it is not possible to obtain a measured height and weight
* People with a definitive diagnosis of dementia
* People who lack capacity to understand the purpose of the study and to consent
* Patients who are unable to understand and speak English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be approached for consideration and recruitment to the study in a stratified manner in order to proportionately represent the diagnostic groups admitted to The Royal Marsden NHS Foundation Trust as inpatients. Patients will be approached sequentially from the list until the required number of patients are recruited for that particular diagnoses. Recruitment for particular diagnostic groups may take place over a number of days until the required number of patients is recruited. The same procedure will be repeated, with a newly generated list, for all selected diagnostic groups in a random order. This methodology will aim to capture patients who have been newly diagnosed, patients with established disease, patients newly admitted and those who have been inpatients for anumber of days or weeks.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Screening Tool | 24 hrs
  The primary endpoint of the study is the sensitivity of each screening tool as compared to the gold standard of PG-SGA when completed by a trained dietitian.

SECONDARY OUTCOMES:
Specificity of the Tool | 24 hrs
  Secondary endpoints are as follows:
  * specificity of the screening tool
  * proportion of inpatients with malnutrition on admission

CONTACTS AND LOCATIONS:
Overall Officials: Clare Shaw, Phd, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, London .., United Kingdom